CLINICAL TRIAL: NCT00199810
Title: Hemodynamic Measurements in Women With Serious Preeclampsia
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Eldrid Langesæter, Consultant, MD, PhD, Oslo University Hospital
Other Study IDs: Elangepreeklampsi2005-; S-05173
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Preeclampsia
Keywords: Cardiac output; Preeclamptic women; systemic vascular resistance; blood pressure
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This trial is examining hemodynamic measurements in women with serious preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Women with serious preeclampsia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with moderate-to-severe pre-eclampsia
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2005-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Hemodynamic variations in preeclamptic women | days

SECONDARY OUTCOMES:
Urine output | days
thrombocyte count | days

CONTACTS AND LOCATIONS:
Overall Officials: Eldrid Langesæter Langesæter, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway